CLINICAL TRIAL: NCT02087761
Title: A Multi-Site Clinical Evaluation of the ARIES Flu Assay in Symptomatic Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Luminex Corporation (Industry)
Responsible Party: Sponsor
Organization: Luminex Molecular Diagnostics (Industry)
Other Study IDs: LMA-FLU-01-CS-001
Record Dates: First submitted 2014-03-12; First posted 2014-03-14 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-03

CONDITIONS: Respiratory Tract Infection; Bronchitis; Pneumonia
Keywords: ARIES Flu
MeSH Terms: conditions — Respiratory Tract Infections; Bronchitis; Pneumonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasal-pharyngeal swabs
Oversight: Data Monitoring Committee: No

SUMMARY:
The ARIES Flu Assay is a real-time PCR based qualitative assay for the direct detection and differentiation of respiratory viral nucleic acid in nasopharyngeal swabs specimens.

The objective of this study is to establish the diagnostic accuracy of ARIES Flu Assay.

DETAILED DESCRIPTION:
The ARIES Flu Assay is a real-time polymerase chain reaction (PCR) based qualitative in vitro diagnostic test for the direct detection and differentiation of respiratory viral nucleic acid in nasopharyngeal swabs specimens from patients with signs and symptoms of respiratory tract infection in conjunction with clinical and laboratory findings.

The objective is to establish the diagnostic accuracy of ARIES Flu Assay through a multi-site, method comparison on prospectively collected, left-over, and de-identified, nasopharyngeal swab specimens. Diagnostic accuracy will be expressed in terms of clinical sensitivity (or positive agreement) and specificity (or negative agreement).

ELIGIBILITY:
Inclusion Criteria:

* The specimen is from a patient suspected of having respiratory tract infection for whom a requisition has been made for viral testing
* The specimen is from a male of female subject who was either hospitalized, admitted to a hospital emergency department or visiting an outpatient clinic.
* The specimen is a nasopharyngeal swab

Exclusion Criteria:

* The specimen is NOT a nasopharyngeal swab
* The specimen was not properly collected, transported or stored according to the instructions provided by the sponsor.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All comers
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy will be expressed in terms of clinical sensitivity (or positive agreement) and specificity (or negative agreement). | Within the first year of sample collection
  Accuracy determinations (diagnostic sensitivity and specificity, positive and negative agreement) were based on the fraction of comparator positive (or negative) results which were also positive (or negative) by ARIES Flu assay.

CONTACTS AND LOCATIONS:
Overall Officials: David Himsworth, Study Director — Luminex Corporation
Locations (3):
- United States (3):
  - St. Louis Children's Hospital, St Louis, Missouri
  - North Shore-LIJ Health System Laboratories, Lake Success, New York
  - Baylor Scott & White Health, Temple, Texas